CLINICAL TRIAL: NCT04999592
Title: Ceftriaxone to PRevent pneumOnia and inflammatTion aftEr Cardiac arresT (PROTECT): a Randomized-controlled Trial and Microbiome Assessment
Brief Title: Ceftriaxone to PRevent pneumOnia and inflammatTion aftEr Cardiac arresT (PROTECT)
Acronym: PROTECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lapse in funding
Sponsor: David J. Gagnon (Other)
Collaborators: MaineHealth (Other); National Institute of General Medical Sciences (NIGMS) (NIH); University of New England (Other)
Responsible Party: Sponsor-Investigator, David J. Gagnon, Critical Care Clinical Pharmacist, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1P20GM139745-01 (NIH); P20GM139745 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-08-11 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Pneumonia
Keywords: out-of-hospital cardiac arrest; cardiac arrest; pneumonia; randomized clinical trial; infection; ceftriaxone; microbiome; inflammation; prophylaxis
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Pneumonia; Heart Arrest; Infections; Inflammation | interventions — Standard of Care; Antibiotic Prophylaxis; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical team responsible for the participant (physicians, nurses and others) and involved with direct patient care will be blinded. Investigators will be blinded and the placebo will match the study drug. Outcomes Assessors will be blinded to treatment assignment during assessments of pneumonia and functional outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- No prophylaxis (placebo) (Active Comparator): Standard care without antibiotic prophylaxis and treatment of infection if clinically warranted.
  Administer antibiotics in response to infection.
  Interventions: Drug: Standard of care without prophylaxis
- Prophylaxis (Experimental): Antibiotic prophylaxis for 3 days. Antibiotic prophylaxis with Ceftriaxone 2 gm IV q12h for 3 days.
  Interventions: Drug: Antibiotic prophylaxis

INTERVENTIONS:
Drug: Standard of care without prophylaxis — Administer antibiotics in response to infection
  Other Names: Placebo
  Arms: No prophylaxis (placebo)
Drug: Antibiotic prophylaxis — Ceftriaxone 2 gm IV q12h for 3 days
  Other Names: Rocephin (ceftriaxone)
  Arms: Prophylaxis

SUMMARY:
Randomized-controlled trial and microbiome assessment to understand the risk-to-benefit ratio of prophylactic antibiotics (Ceftriaxone) vs placebo in patients with pneumonia and inflammation after cardiac arrest outside the hospital.

DETAILED DESCRIPTION:
Pneumonia is an infection of the lungs resulting in alveolar inflammation and fluid or purulent material accumulation. It is the most common infection after cardiac arrest occurring in up to 65% of patients treated with targeted temperature management. Pneumonia may result from aspiration during cardiopulmonary resuscitation (CPR), or by introduction of oropharyngeal flora into the lungs during airway management. Preventing infection after OHCA may: 1) reduce exposure to broad-spectrum antibiotics and subsequent collateral damage, 2) prevent hemodynamic derangements due to local and systemic inflammation, and 3) prevent an association between infection and morbidity and mortality. These benefits must be balanced with the risk for altering bacterial resistomes in the absence clinical infection. Accordingly, further study is warranted to understand the risk-to-benefit ratio of prophylactic antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Comatose (do not follow simple verbal commands)
* Have any initial heart rhythm (shockable or non-shockable)
* OHCA including the emergency department

Exclusion Criteria:

* Name on opt-out list
* In-hospital cardiac arrest
* Interval >6 hours from ICU admission to study drug receipt
* Preexisting terminal disease making 180-day survival unlikely
* Refused informed consent
* Emergent coronary artery bypass grafting
* Anaphylaxis or angioedema to beta-lactam antibiotics (i.e., cephalosporins or penicillins)
* Under legal guardianship or prisoner
* Known colonization with methicillin-resistant Staphylococcus aureus (MRSA) or vancomycin-resistant enterococcus (VRE)
* Clinical bacterial infection prior to hospital admission defined as any one of the following:

  * Infectious prodrome preceding OHCA
  * Active course of antibiotics for infection prior to admission
  * Active infection documented in the electronic medical record
  * Family or surrogate endorsement of an active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gagnon, PharmD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gagnon DJ, Ryzhov SV, May MA, Riker RR, Geller B, May TL, Bockian S, deKay JT, Eldridge A, Van der Kloot T, Lerwick P, Lord C, Lucas FL, Mailloux P, McCrum B, Searight M, Wirth J, Zuckerman J, Sawyer D, Seder DB. Ceftriaxone to PRevent pneumOnia and inflammaTion aftEr Cardiac arresT (PROTECT): study protocol for a randomized, placebo-controlled trial. Trials. 2022 Mar 4;23(1):197. doi: 10.1186/s13063-022-06127-w. PMID 35246202
- [Derived] Gagnon DJ, Burkholder KM, Weissman AJ, Riker RR, Ryzhov S, May TL, DiPalazzo J, deKay JT, Knudsen L, Moore MW, Pozzessere NA, Weatherbee M, Kelly M, Nigatu AS, Sevigny JL, Simpson S, Thomas WK, Callaway CW, Geller BJ, Sawyer DB, Seder DB. Ceftriaxone to Prevent Early-Onset Pneumonia in Comatose Patients Following Out-of-Hospital Cardiac Arrest: A Pilot Randomized Controlled Trial and Resistome Assessment (PROTECT). Chest. 2026 Jan;169(1):115-127. doi: 10.1016/j.chest.2025.08.007. Epub 2025 Aug 28. PMID 40885534

RESULTS

PARTICIPANT FLOW:
Groups:
- No Prophylaxis (Placebo): Standard care without antibiotic prophylaxis and treatment of infection if clinically warranted.
  Administer antibiotics in response to infection.
  Standard of care without prophylaxis: Administer antibiotics in response to infection
Period: Overall Study
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Started | 27 | 26
Completed | 26 | 26
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 53 subjects were consented and 1 withdrew consent leaving 52 subjects (26 in each arm) evaluable.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [52 to 65] | 60 [52 to 67] | 60 [52 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 25 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 25 | 50
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinically-diagnosed Early-onset Pneumonia
Description: Percentage of Participants with Clinically-diagnosed Early-onset Pneumonia occurring <4 days after initiation of mechanical ventilation
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 18 | 10

2. Secondary Outcome: Microbiologically-confirmed Early-onset Pneumonia
Description: Percentage of Participants with Microbiologically-confirmed Early-onset Pneumonia occurring <4 days after initiation of mechanical ventilation
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 13 | 6

3. Secondary Outcome: Microbiologically-confirmed Late-onset Pneumonia
Description: Percentage of Participants with Microbiologically-confirmed late-onset pneumonia occurring ≥4 days after initiation of mechanical ventilation
Time Frame: ≥ 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 4 | 1

4. Secondary Outcome: Clinically-diagnosed Late-onset Pneumonia
Description: Percentage of Participants with Clinically-diagnosed late-onset pneumonia occurring ≥4 days after initiation of mechanical ventilation
Time Frame: ≥ 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 6 | 3

5. Secondary Outcome: Non-pulmonary Infections
Description: Percentage of Participants with non-pulmonary infections
Time Frame: During the intervention and immediately after the intervention until hospital discharge, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 0 | 0

6. Secondary Outcome: ICU-free Days During Admission
Description: ICU-free days in the first 28 days of admission
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
days | 0 [0 to 2] | 16 [0 to 24]

7. Secondary Outcome: Mechanical Ventilator-free Days During Admission
Description: Mechanical ventilator-free days in the first 28 days of admission
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
days | 0 [0 to 8] | 25 [0 to 26]

8. Secondary Outcome: Death in the Hospital
Description: Percentage of Participants who Die in the Hospital during admission
Time Frame: During the intervention (3 days) and immediately after the intervention until subject death or hospital discharge, an average of 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 19 | 11

9. Secondary Outcome: Functional Outcome at 6 Months Post-hospital Discharge
Description: Median mRS (0 as no residual symptoms and 6 as death) at 6 Months Post-hospital Discharge
Time Frame: 6 months post-hospital discharge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
units on a scale | 6 [6 to 6] | 6 [1 to 6]

10. Secondary Outcome: Clostridioides Difficile-associated Diarrhea
Description: Percentage of Participants with Clostridioides difficile-associated Diarrhea
Time Frame: During the intervention and immediately after the intervention until death or hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 0 | 0

11. Secondary Outcome: Type One Hypersensitivity Reactions
Description: Percentage of Participants with Type One (immediate-type) hypersensitivity reactions
Time Frame: Three days
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 0 | 0

12. Secondary Outcome: Participants With Gallbladder Disease
Description: Percentage of Participants with Gallbladder disease
Time Frame: During the intervention and immediately after the intervention until death or hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
Number analyzed (Participants) | 26 | 26
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment to hospital discharge or death, whichever occurred first, on average 30 days
Arm/Group | No Prophylaxis (Placebo) | Prophylaxis
All-Cause Mortality (participants affected / at risk) | 19/26 | 11/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT04999592/Prot_SAP_000.pdf